CLINICAL TRIAL: NCT05530967
Title: Assessing the Structure and Validity of the PAP Problems Triage Tool in Patients With Newly-Initiated PAP Treatment for Obstructive Sleep Apnea
Brief Title: Assessing the Validity of the PAP Problems Triage Tool in Patients With PAP Treatment for Obstructive Sleep Apnea
Acronym: TriagingTool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Dennis Hwang, MD, Medical Director, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KPSleep-006
Record Dates: First submitted 2022-07-05; First posted 2022-09-07 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Positive Airway Pressure (PAP) Therapy; Triaging Tool; PAP Problems; PAP Adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triaging Tool (Experimental)
  Interventions: Other: TT
- Video Education (Experimental)
  Interventions: Other: TT; Other: VE

INTERVENTIONS:
Other: TT — This intervention uses questionnaire at three-time intervals (i.e., days 5, 10, and 30) and abstraction of PAP use data (days 1 - 35). Consecutive adults with moderate-severe OSA and recommended to PAP treatment will be invited to the study. Once the patient has been prescribed PAP therapy a research associate will call the patient before receiving their new PAP device. The research associate will utilize an IRB approved telephone script to discuss study details, conduct eligibility screening (inclusion/exclusion criteria), and to ask whether the patient is interested in participating.
  The research associate will then send the patient an IRB approved digital information sheet. The information sheet will provide the patient an option to mark "Yes" if they are willing to participate in the study or "No" if they are not willing. Patients who indicate their willingness to participate will receive the Triage Tool in accordance with the study protocol.
Other: VE — A randomly selected sub-group of participants (n=30) will also receive an animated education video that provides targeted information and encouragement for self-managing your PAP problem(s). Patients in this sub-group will be asked to view a maximum of 2 different videos that are less than 2 minutes in duration. These videos are aligned with practice guideline recommendations for addressing PAP problems early in treatment. The videos will be sent digitally from Somnoware™.
  Arms: Video Education

SUMMARY:
The intended use of the Positive Airway Pressure (PAP) Problems Triaging Tool (TT) is to appropriately triage patients with a PAP-associated problem(s) to a specific intervention(s) based on patient responses. Thus, the proposed research will validate the tool, determine optimal scoring thresholds, and explore the utility of the tool as an indicator for intervention. Our central hypothesis is that the PAP Problems TT will identify treatment barriers that if unaddressed, are predictive of treatment non-adherence.

DETAILED DESCRIPTION:
This study is a one-group observational design that uses a TT questionnaire and abstraction of PAP use data from a clinically available interface (Somnoware™). Consecutive adults with OSA and recommended to PAP treatment at the Fontana Medical Sleep Center will be invited to the study. Once the patient has been prescribed PAP therapy and has indicated their willingness to participate the TT will be sent digitally from Somnoware™. Participants will receive the TT in accordance to the next time interval defined by the study protocol. A randomly selected sub-group of participants will automatically receive an animated education video delivered digitally from Somnoware™. These videos will provide targeted information for self-managing the endorsed PAP problem.

Diagnostic polysomnogram (PSG) or home sleep apnea test (HSAT) data will be abstracted from Somnoware™. Daily PAP data will be abstracted from Somnoware™ for the first 35-days of PAP use. Demographic data will also be abstracted at day 35 (from the patient's clinical intake questionnaire and electronic health record).

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Member (KP insured)
* OSA diagnosis by polysomnogram or Home Sleep Apnea Test with Apnea Hypopnea Index ≥ 15 events/hour
* PAP naïve
* Able to consent to participate
* Fluent or proficient with English
* Accepts PAP for home treatment

Exclusion Criteria:

* Chronic respiratory failure requiring Oxygen supplementation
* PAP device other than a PAP or AutoPAP (i.e., bilevel PAP)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Factor Analysis | 30 days
  Investigate the factor structure of the TT, an exploratory factor analysis (EFA) will be conducted. A forced six-factor EFA using a varimax rotation will be conducted to determine the factor loadings on six sub-scales and to determine whether the EFA factors are similar to the theoretically derived categories from the original TT instrument. Data from the TT collected at day 5 will be used for the factor analysis as we expect higher response rate at this first data collection endpo
Triaging Tool Validity | 30 days
  Concurrent validity will assess the extent to which TT scores are related to concurrent PAP use. This will be established based on Pearson product moment correlation coefficients (for continuous PAP use [hours/night]) and Point Biserial correlations (for PAP non-adherence, defined as <4 hours/night of use, on average) at three intervals: day 5 (PAP use on days 1-5), day 10 (PAP use on days 6-10), and day 30 (PAP use on days 11-30).
Triaging Tool Predictive Validity | 30 days
  To determine the TT accuracy for predicting PAP non-adherence (defined as <4 hours/night of use, on average) receiver operating characteristic (ROC) curves and respective area under the curve (AUC) with 95% confidence interval (CI) will be estimated using PAP TT subdomain scores as predictors for PAP non-adherence within 5 days post-TT score data collection. As TT data will be collected at 3 intervals (i.e., days 5, 10, and 30) and considering the 6 subdomains from the TT scale, a total of 18 ROCs/AUCs will be estimated.

SECONDARY OUTCOMES:
Changes in PAP Use Utilizing Video Education | 5 days
  Unadjusted, descriptive analysis will be conducted to explore acute changes in PAP use immediately after intervention delivery. Change in PAP use will be assessed by computing the difference (delta) in PAP use (mean, hours/night) for the 5 consecutive days pre- and post-VE. Positive delta values will indicate greater PAP use post-intervention delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No